CLINICAL TRIAL: NCT00510068
Title: A Randomized Double-blind Phase III Study of RAD001 10 mg/d Plus Best Supportive Care Versus Placebo Plus Best Supportive Care in the Treatment of Patients With Advanced Pancreatic Neuroendocrine Tumor (NET)
Brief Title: Efficacy and Safety of Everolimus (RAD001) Compared to Placebo in Patients With Advanced Neuroendocrine Tumors
Acronym: RADIANT-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001C2324; 2006-006819-75 (EudraCT Number)
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Results first posted 2011-12-15 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Advanced Neuroendocrine Tumors of Pancreatic Origin
Keywords: Phase III; Advanced Neuroendocrine Tumor in adults; RAD001; NET; everolimus; mTOr; islet cell; neuroendocrine
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus 10 mg/day (Experimental): Participants received 10 mg per day of Everolimus plus best supportive care. Patients received their first dose of everolimus at Visit 2 (Cycle 1 Day 1).
  Interventions: Drug: Everolimus
- Placebo (Placebo Comparator): Participants received matching placebo to everolimus daily plus best supportive care. Patients received their first dose of matching placebo at Visit 2 (Cycle 1 Day 1).
  Interventions: Drug: Everolimus Placebo

INTERVENTIONS:
Drug: Everolimus — A 10-mg dose of everolimus was given by continuous oral daily dosing of two 5-mg tablets.
  Other Names: RAD001
  Arms: Everolimus 10 mg/day
Drug: Everolimus Placebo — a 10-mg dose of matching placebo to Everolimus was given by continuous oral daily dosing of two 5-mg tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate progression free survival in those participants assigned everolimus 10 mg/day plus Best Supportive Care versus those assigned to placebo plus Best Supportive Care in Advanced Neuroendocrine Tumors of pancreatic origin.

ELIGIBILITY:
Inclusion criteria:

1. Patients must have advanced (unresectable or metastatic) biopsy-proven pancreatic NET
2. Measurable disease by radiologic assessment
3. Adequate blood work
4. Performance Status 0-2 : Ability to be out of bed most of the time
5. Adult male or female patients ≥ 18 years of age
6. Women of childbearing potential must have a negative serum pregnancy test
7. Written informed consent from patients must be obtained in accordance to local guidelines

Exclusion criteria:

1. Patients with severe kind of (poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid and small cell carcinoma) cancer are not eligible
2. Other chemotherapy, immunotherapy or radiotherapy within 4 weeks prior to starting this trial
3. Hepatic artery procedure called embolization within the last 6 months (1 month if there are other sites of measurable disease), or cryoablation/ radiofrequency ablation of hepatic metastasis within 2 months of enrollment
4. Prior therapy with the same kind of medication (mTOR inhibitors: sirolimus, temsirolimus, everolimus).
5. Uncontrolled diabetes mellitus Patients who have any severe and/or uncontrolled medical conditions such as:
6. Patients receiving chronic treatment with corticosteroids or another immunosuppressive agent
7. Patients with a known history of HIV seropositivity
8. No other prior or concurrent cancer at the time enrolling to this trial

Other protocol defined inclusion/ exclusion criteria applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (74):
- United States (24):
  - University of South Alabama / Mitchell Cancer Institute Deptof Mitchell Cancer Inst(2), Mobile, Alabama
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Cedars Sinai Medical Center SC-2, Los Angeles, California
  - University of California at Los Angeles UCLA (3), Los Angeles, California
  - University of California San Francisco Dept. of UCSF Comp. Cancer, San Francisco, California
  - Kaiser Permanente Northwest Franklin Medical Offices, Denver, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute Malignant Hematology Clinic, Tampa, Florida
  - Indiana University Health Goshen Center for Cancer Dept. of Indiana Univ. Cancer, Indianapolis, Indiana
  - University of Iowa Medical Center Dept. of Iowa Medical Center, Iowa City, Iowa
  - University of Louisville / James Graham Brown Cancer Center SC, Louisville, Kentucky
  - LSU HEALTH SCIENCES CENTER/ LSU SCHOOL OF MEDICINE Dept. of Neuroendocrine Clinic, New Orleans, Louisiana
  - Boston Medical Center BMC, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute Dept.of KarmanosCancerInst (4), Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Littleton Regional Hospital Dept. of Hematology/Oncology, Littleton, New Hampshire
  - Columbia University Medical Center- New York Presbyterian Dept. of Columbia Med. Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Ohio State Comprehensive Cancer Center/James Cancer Hospital Dept. of OHSU Medical Center, Columbus, Ohio
  - Oregon Health & Science University Dept. of OHSU (3), Portland, Oregon
  - St. Luke's Hospital and Health Network St. Luke's Cancer Network, Bethlehem, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - University of Texas/MD Anderson Cancer Center Dept of MD Anderson CancerCent, Houston, Texas
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Fortaleza, Ceará, Brazil
- Canada (4):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (12):
  - Novartis Investigative Site, Strasbourg, France
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (5):
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
- Italy (4):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pisa, PI
- Japan (3):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Chuo-ku, Tokyo
- Novartis Investigative Site, Groningen, Netherlands
- Novartis Investigative Site, Martin, Slovak Republic, Slovakia
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
- Novartis Investigative Site, Uppsala, Sweden
- Novartis Investigative Site, Zurich, Switzerland, Switzerland
- Taiwan (4):
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Lin-Ko
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla
- United Kingdom (3):
  - Novartis Investigative Site, Withington, Greater Manchester
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

REFERENCES:
- [Derived] Chan DL, Yao JC, Carnaghi C, Buzzoni R, Herbst F, Ridolfi A, Strosberg J, Kulke MH, Pavel M, Singh S. Markers of Systemic Inflammation in Neuroendocrine Tumors: A Pooled Analysis of the RADIANT-3 and RADIANT-4 Studies. Pancreas. 2021 Feb 1;50(2):130-137. doi: 10.1097/MPA.0000000000001745. PMID 33560090
- [Derived] Yao JC, Voi M, Lincy J, Pavel M. Reply to V. Amoroso et al. J Clin Oncol. 2017 May 1;35(13):1488-1489. doi: 10.1200/JCO.2017.71.3875. Epub 2017 Jan 23. No abstract available. PMID 28113028
- [Derived] Yao JC, Pavel M, Lombard-Bohas C, Van Cutsem E, Voi M, Brandt U, He W, Chen D, Capdevila J, de Vries EGE, Tomassetti P, Hobday T, Pommier R, Oberg K. Everolimus for the Treatment of Advanced Pancreatic Neuroendocrine Tumors: Overall Survival and Circulating Biomarkers From the Randomized, Phase III RADIANT-3 Study. J Clin Oncol. 2016 Nov 10;34(32):3906-3913. doi: 10.1200/JCO.2016.68.0702. Epub 2016 Sep 30. PMID 27621394
- [Derived] Lombard-Bohas C, Yao JC, Hobday T, Van Cutsem E, Wolin EM, Panneerselvam A, Stergiopoulos S, Shah MH, Capdevila J, Pommier R. Impact of prior chemotherapy use on the efficacy of everolimus in patients with advanced pancreatic neuroendocrine tumors: a subgroup analysis of the phase III RADIANT-3 trial. Pancreas. 2015 Mar;44(2):181-9. doi: 10.1097/MPA.0000000000000262. PMID 25479584
- [Derived] Yao JC, Shah MH, Ito T, Bohas CL, Wolin EM, Van Cutsem E, Hobday TJ, Okusaka T, Capdevila J, de Vries EG, Tomassetti P, Pavel ME, Hoosen S, Haas T, Lincy J, Lebwohl D, Oberg K; RAD001 in Advanced Neuroendocrine Tumors, Third Trial (RADIANT-3) Study Group. Everolimus for advanced pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):514-23. doi: 10.1056/NEJMoa1009290. PMID 21306238

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Period
Arm/Group | Everolimus 10 mg/Day | Placebo
Started | 207 | 203
Safety Population | 204 | 203
Completed | 0 | 0
Not Completed | 207 | 203
Not completed — Disease progression | 98 | 169
Not completed — Final primary analysis | 52 | 18
Not completed — Adverse Event | 37 | 7
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Death | 4 | 3
Not completed — Abnormal test result (s) | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 6 | 0
Period: Open-label Period
Arm/Group | Everolimus 10 mg/Day | Placebo
Started | 225 (172 patients switched over from placebo & 53 who were initially randomized to Everolimus arm.) | 0
Completed | 0 | 0
Not Completed | 225 | 0
Not completed — Disease Progression | 124 | 0
Not completed — Adverse Event | 46 | 0
Not completed — Withdrawal by Subject | 21 | 0
Not completed — Administrative problems | 17 | 0
Not completed — Death | 7 | 0
Not completed — New cancer therapy | 7 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Abnormal laboratory value (s) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus 10 mg/Day | Placebo | Total
Number analyzed (Participants) | 207 | 203 | 410
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (12.2) | 56.2 (11.4) | 56.6 (11.8)
Age, Customized [Number; unit: Participants]
  <65 years | 146 | 153 | 299
  >=65 years | 61 | 50 | 111
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 86 | 183
  Male | 110 | 117 | 227
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 156 | 166 | 322
  Asian | 40 | 34 | 74
  Black | 9 | 2 | 11
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression Free Survival (PFS) Based as Per Investigator Using Kaplan-Meier Methodology
Description: Progression of disease is defined as the time from study start to the date of first documented progression of disease or death due to any cause. Progression of disease is defined by RECIST criteria: Progression = 20% increase in the sum of the longest diameter of all target lesions, from the smallest sum of longest diameter of all target lesions recorded at or after baseline; or a new lesion; or progression of non-target lesions.
Time Frame: Time from randomisation to dates of disease progression, death from any cause or last tumor assessment, reported between day of first patient randomised, 17 August 2007, until cut-off date 28 February 2010
Population: The Full Analysis Set (FAS) consists of all patients who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
Months | 11.04 [8.41 to 13.86] | 4.60 [3.06 to 5.39]

2. Secondary Outcome: Percentage of Participants With Objective Response Rate ( CR {Complete Response} OR PR {Partial Response})
Description: Objective Response defined by RECIST criteria: Partial response (PR) must have ≥ 30% decrease in the sum of the longest diameter of all target lesions, from the baseline sum. Complete response (CR) must have disappearance of all target and non-target lesions. For CR or PR, tumor measurements must be confirmed by 2nd assessments within 4 weeks . Progression = 20% increase in the sum of the longest diameter of all target lesions, from the smallest sum of longest diameter of all target lesions recorded at or after baseline; or a new lesion; or progression of non-target lesions
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) consists of all patients who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
Percentage of participants | 4.8 [2.3 to 8.7] | 2.0 [0.5 to 5.0]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from date of randomization to the date of death due to any cause. Analyses were performed using all deaths in the FAS population regardless of whether they were observed during the double-blind treatment period, the open-label treatment period, the post-treatment evaluations, or the survival follow-up period.
Time Frame: Baseline, to death- no time limit
Population: The Full Analysis Set (FAS) included all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
Months | 44.02 [35.61 to 51.75] | 37.68 [29.14 to 45.77]

4. Secondary Outcome: Progression Free Survival According to Ki-67 Levels Categorized as: Less Than or Equal to 2%, > 2% to Less Than or Equal to 5% and > 5%
Description: The level of Ki 67 expression for evaluable tumor samples were analyzed towards progression free survival (PFS) as per local investigator assessment. The Ki-67 protein is a cellular marker for proliferation. It is strictly associated with cell proliferation. During interphase, the Ki-67 antigen can be exclusively detected within the cell nucleus, whereas in mitosis most of the protein is relocated to the surface of the chromosomes. Baseline Ki 67 levels were categorized as: less than or equal to 2%, > 2% to less than or equal to 5% and > 5%.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) consisted of all patients who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
Months
  Ki67 <=2% (n: 7, 17) | 12.52 [3.42 to 14.75] | 3.68 [2.86 to 5.52]
  2% <Ki67 <=5% (n: 24, 13) | 10.94 [5.55 to 16.59] | 8.48 [3.78 to 13.83]
  Ki67 >5% (n: 20, 22) | 7.69 [5.59 to NA] — Upper boundary of the 95% (Confidence Interval (CI) was not computable | 3.15 [2.79 to 5.55]

5. Secondary Outcome: Progression Free Survival According to Chromogramin A Tumor Marker (CgA) Baseline Level and According to CgA Early Response
Description: Baseline levels of serum CgA SE were characterized towards progression free survival (PFS) as per local investigator assessment, relative to the upper limited of normal (ULN). CgA levels exceeding 2 x ULN were considered to be 'Elevated' otherwise considered as "Non-elevated". An 'early response' (applicable to only those patients with elevated levels at baseline) was defined as a decrease of greater than or equal to 30% from baseline to Cycle 2 Day 1 or normalization by Cycle 2 Day 1. CgA is widely expressed in well-differentiated pancreatic NET. CgA is present in the secretory granules of neuroendocrine cells. Pancreatic NET patients often present with elevated circulating levels of CgA in their blood. Baseline levels of these biomarkers are considered as prognostic factors.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) consisted of all patients who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
Months
  CgA Levels at baseline: CgA <= 2x ULN (n:121, 97) | 11.17 [8.54 to 16.49] | 4.90 [2.99 to 5.55]
  CgA levels at baseline: CgA > 2x ULN (n:84, 103) | 8.54 [7.69 to 13.80] | 4.34 [2.86 to 5.39]
  Early CgA response: Response (n: 48, 22) | 8.54 [7.56 to 14.00] | 5.70 [3.19 to 8.54]
  Early CgA response: Non-Response (n:40, 82) | 11.14 [6.90 to NA] — Upper boundary of the 95% Confidence Interval (CI) was not be computable | 3.19 [2.83 to 5.36]

6. Secondary Outcome: Progression Free Survival According to Neuron Specific Enolase Tumor Marker (NSE) Baseline Level and According to NSE Early Response
Description: Baseline levels of serum NSE were characterized towards PFS as per local investigator assessment, relative to the upper limited of normal (ULN). NSE levels exceeding ULN were considered to be 'Elevated' otherwise considered as "Non-elevated". An 'early response' (applicable to only those patients with elevated levels at baseline) was defined as a decrease of greater than or equal to 30% from baseline to Cycle 2 Day 1 or normalization by Cycle 2 Day 1. NSE is widely expressed in well-differentiated pancreatic NET. NSE is usually expressed in the cytoplasm. Pancreatic NET patients often present with elevated circulating levels of NSE in their blood. Baseline levels of these biomarkers are considered as prognostic factors.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) consisted of all patients who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
Months
  NSE Levels at baseline: <= ULN (n: 155, 138) | 13.86 [10.81 to 18.10] | 5.36 [3.78 to 5.55]
  NSE levels at baseline: > ULN (n: 48, 56) | 8.11 [4.24 to 11.17] | 2.83 [2.60 to 3.06]
  Early NSE response: Response (n: 24, 16) | 8.11 [4.24 to 11.40] | 3.06 [2.23 to 5.36]
  Early NSE response: Non-Response (n:16, 27) | 3.79 [2.60 to 13.80] | 2.58 [1.84 to 2.83]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs)
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: on or after the start of double-blind study medication until no later than 28 days after double-blind study medication discontinuation
Population: The Safety Set consists of all patients who received any study drug and had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 204 | 203
Participants
  Adverse events (AEs) | 203 | 198
  Death | 111 | 23
  Serious Adverse Events | 84 | 52

8. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) (Open-label Period)
Description: as for outcome 7
Time Frame: on or after the start of open-label study medication until no later than 28 days after open-label study medication discontinuation
Population: The open-label set was used to summarize the safety analyses performed on data collected in the open-label period of the study: the open-label set included only patients who received at least one dose of open-label everolimus 10 mg and had at least one safety assessment during the open-label period of the study.
Measure: Number; unit: Participants
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 225 | 0
Participants
  Adverse events (AEs) | 221 |
  Death | 122 |
  Serious Adverse Events | 108 |

9. Secondary Outcome: Evaluation of Pharmacokinetics (PK) Parameter: AUC0-t Last
Description: The PK parameters for a full PK profile at steady-state were determined in blood using non compartmental methods. This PK parameter is area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-t last).
Time Frame: Day 1 of every cycle (28 days/cycle) throughout the study
Population: The Safety Set consisted of all patients who received any study drug and had at least one postbaseline safety assessment.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Groups:
- Everolimus 5 mg/Day: Participants received 5 mg per day of everolimus plus best supportive care. Patients received their first dose of everolimus at Visit 2 (Cycle 1 Day 1).
Arm/Group | Everolimus 10 mg/Day | Everolimus 5 mg/Day
Number analyzed (Participants) | 7 | 1
ng.h/mL | 594 (313) | 481 (NA) — Summary statistics were only produced if the sample size for the dose group in the respective cycle is 3 or more.

10. Secondary Outcome: Evaluation of Pharmacokinetics (PK) Parameters: Cmax, Cmin
Description: The PK parameters for a full PK profile at steady-state were determined in blood using non compartmental methods. The PK parameter: maximum (peak) drug concentration (Cmax) and minimum (trough) drug concentration (Cmin).
Time Frame: Day 1 of every cycle (28 days/cycle) throughout the study
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus 10 mg/Day | Everolimus 5 mg/Day
Number analyzed (Participants) | 7 | 1
ng/mL
  Cmax | 62.4 (18.5) | 27.4 (NA) — Summary statistics will only be produced if the sample size for the dose group in the respective cycle is 3 or more.
  Cmin | 9.80 (4.95) | 12.2 (NA) — Summary statistics will only be produced if the sample size for the dose group in the respective cycle is 3 or more.

11. Secondary Outcome: Evaluation of Pharmacokinetics (PK) Parameter: CL/F
Description: The PK parameters for a full PK profile at steady-state were determined in blood using non compartmental methods. The PK parameter clearance of distribution expressed as a function of bioavailability (CL/F).
Time Frame: Day 1 of every cycle (28 days/cycle) throughout the study
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Everolimus 10 mg/Day | Everolimus 5 mg/Day
Number analyzed (Participants) | 7 | 1
L/h | 20.2 (7.7) | 10.7 (NA) — Summary statistics were only produced if the sample size for the dose group in the respective cycle is 3 or more.

12. Secondary Outcome: Evaluation of Pharmacokinetics (PK) Parameter: Tmax -Time to Maximum (Peak) Drug Concentration
Description: The PK parameters for a full PK profile at steady-state were determined in blood using non compartmental methods. Values for tmax where summarized in median (range).
Time Frame: Day 1 of every cycle (28 days/cycle) throughout the study
Population: as for outcome 9
Measure: Median (Full Range); unit: h
Arm/Group | Everolimus 10 mg/Day | Everolimus 5 mg/Day
Number analyzed (Participants) | 7 | 1
h | 1.17 [0.5 to 24.0] | 3.0 [NA to NA] — Summary statistics were only produced if the sample size for the dose group in the respective cycle is 3 or more.

13. Secondary Outcome: Analysis of Time to Definitive Deterioration of WHO Performance Status Using Kaplan-Meier
Description: Time to definitive worsening is defined as a definitive increase in performance status from a baseline of 0 or 1 to WHO >= 2, or from a baseline value of 2 to WHO >= 3. If no earlier deterioration, patients were censored at the end of follow-up or at the start of further antineoplastic therapy. Rates of patients with no deterioration at 3 and 6 months were computed using Kaplan-meier method. Grade 0: Able to carry out all activity without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to do light work; Grade 2: Ambulatory & capable of all self-care but unable to carry out any work. Up & about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled & cannot carry on any self-care; totally confined to bed or chair.
Time Frame: 3 months, 6 months
Population: The Full Analysis Set (FAS) consists of all patients who were randomized.
Measure: Number; unit: % of participants with no deterioration
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
% of participants with no deterioration
  Month 3 | 94.4 [90.0 to 96.8] | 91.8 [86.8 to 95.0]
  Month 6 | 90.6 [85.2 to 94.0] | 86.3 [79.3 to 91.0]

14. Secondary Outcome: Plasma Angiogenesis Marker: Basic Fibroblast Growth Factor (bFGF)
Description: This biomarker is related to angiogenesis pathway, was analyzed to determine the effects of everolimus on plasma antiangiogenic molecules.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1
Population: The Full Analysis Set (FAS) consists of all patients who were randomized.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
pg/mL
  Baseline (n:198, 195) | 52.59 (101.659) | 51.49 (78.049)
  Cycle 2 Day 1 (n: 185, 184) | 38.43 (51.809) | 58.33 (72.938)
  Cycle 3 Day 1 (n: 185, 174) | 51.97 (89.064) | 59.08 (72.495)
  Cycle 4 Day 1 (n: 171, 159) | 51.28 (82.139) | 54.58 (75.350)

15. Secondary Outcome: Plasma Angiogenesis Marker: Placental Growth Factor (PLGF)
Description: as for outcome 14
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1
Population: The Full Analysis Set (FAS) consists of all patients who were randomized.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
pg/mL
  Baseline (n:198, 195) | 45.82 (282.084) | 32.92 (52.586)
  Cycle 2 Day 1 (n: 185, 184) | 25.78 (33.420) | 35.38 (57.135)
  Cycle 3 Day 1 (n: 185, 174) | 26.55 (28.839) | 33.84 (65.361)
  Cycle 4 Day 1 (n: 171, 159) | 25.69 (18.312) | 35.47 (67.314)

16. Secondary Outcome: Plasma Angiogenesis Marker: Soluble Vascular Endothelial Growth Factor Receptor 1 (sVEGFR1)
Description: as for outcome 14
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1
Population: The Full Analysis Set (FAS) consists of all patients who were randomized.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
pg/mL
  Baseline (n:198, 195) | 264.18 (272.190) | 256.69 (187.866)
  Cycle 2 Day 1 (n: 185, 184) | 307.46 (808.316) | 299.03 (541.933)
  Cycle 3 Day 1 (n: 185, 174) | 263.81 (187.329) | 253.37 (250.841)
  Cycle 4 Day 1 (n: 171, 159) | 258.03 (223.980) | 242.17 (163.561)

17. Secondary Outcome: Plasma Angiogenesis Marker: Soluble Vascular Endothelial Growth Factor Receptor 2 (sVEGFR2)
Description: as for outcome 14
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1
Population: The Full Analysis Set (FAS) consists of all patients who were randomized.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
pg/mL
  Baseline (n:197, 193) | 30061.30 (8607.379) | 31299.61 (9091.460)
  Cycle 2 Day 1 (n: 185, 183) | 22691.18 (6793.409) | 30223.21 (8447.992)
  Cycle 3 Day 1 (n: 185, 173) | 22021.23 (6393.414) | 29264.67 (8408.405)
  Cycle 4 Day 1 (n: 172, 158) | 21218.17 (6249.977) | 28308.58 (8477.049)

18. Secondary Outcome: Plasma Angiogenesis Marker: Vascular Endothelial Growth Factor (VEGF)
Description: as for outcome 14
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1
Population: The Full Analysis Set (FAS) consists of all patients who were randomized.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Everolimus 10 mg/Day | Placebo
Number analyzed (Participants) | 207 | 203
pg/mL
  Baseline (n:198, 195) | 265.09 (283.123) | 326.16 (323.891)
  Cycle 2 Day 1 (n: 185, 184) | 243.03 (183.010) | 326.78 (377.752)
  Cycle 3 Day 1 (n: 185, 174) | 280.18 (268.582) | 292.27 (286.154)
  Cycle 4 Day 1 (n: 171, 159) | 283.51 (326.634) | 319.60 (325.409)

ADVERSE EVENTS:
Groups:
- Everolimus 10mg/Day: Afinitor DB: Participants received 10 mg per day of everolimus plus best supportive care. Patients received their first dose of everolimus at Visit 2 (Cycle 1 Day 1).
- Open Label - Everolimus 10mg: Afinitor OL (for data collected in the open-label period of the study): The open-label set included only patients who received at least one dose of open-label everolimus 10 mg and had at least one safety assessment during the open-label period of the study.
Arm/Group | Everolimus 10mg/Day | Placebo | Open Label - Everolimus 10mg
Serious Adverse Events (participants affected / at risk) | 84/204 | 52/203 | 108/225
Other Adverse Events (participants affected / at risk) | 201/204 | 190/203 | 218/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10mg/Day (N=204) | Placebo (N=203) | Open Label - Everolimus 10mg (N=225)
Anaemia (Blood and lymphatic system disorders) | 7 | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 3
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Branchial cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 0 | 1
Ophthalmoplegia (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 5 | 13
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 3
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 3 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 3
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 7
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4 | 10
Asthenia (General disorders) | 5 | 2 | 6
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1
Device occlusion (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 1
General physical health deterioration (General disorders) | 1 | 1 | 3
Generalised oedema (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 8 | 3 | 8
Sudden death (General disorders) | 0 | 0 | 1
Thrombosis in device (General disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 0 | 5
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 3
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 3 | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0 | 2
Lobar pneumonia (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 2
Perihepatic abscess (Infections and infestations) | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2 | 10
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Ammonia increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 5 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Gastrinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic neuroendocrine tumour metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 3
Depressed level of consciousness (Nervous system disorders) | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Epiduritis (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 2
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 3 | 2
Listless (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 3 | 4
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aneurysm ruptured (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10mg/Day (N=204) | Placebo (N=203) | Open Label - Everolimus 10mg (N=225)
Anaemia (Blood and lymphatic system disorders) | 48 | 18 | 55
Leukopenia (Blood and lymphatic system disorders) | 12 | 4 | 9
Lymphopenia (Blood and lymphatic system disorders) | 15 | 6 | 10
Neutropenia (Blood and lymphatic system disorders) | 14 | 4 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 29 | 2 | 20
Abdominal distension (Gastrointestinal disorders) | 18 | 14 | 19
Abdominal pain (Gastrointestinal disorders) | 47 | 48 | 55
Abdominal pain upper (Gastrointestinal disorders) | 30 | 15 | 29
Aphthous stomatitis (Gastrointestinal disorders) | 25 | 8 | 22
Ascites (Gastrointestinal disorders) | 13 | 4 | 7
Constipation (Gastrointestinal disorders) | 30 | 26 | 32
Diarrhoea (Gastrointestinal disorders) | 97 | 47 | 96
Dry mouth (Gastrointestinal disorders) | 23 | 9 | 8
Dyspepsia (Gastrointestinal disorders) | 13 | 13 | 8
Flatulence (Gastrointestinal disorders) | 10 | 8 | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 6 | 13
Haemorrhoids (Gastrointestinal disorders) | 6 | 4 | 17
Mouth ulceration (Gastrointestinal disorders) | 14 | 4 | 15
Nausea (Gastrointestinal disorders) | 66 | 64 | 80
Stomatitis (Gastrointestinal disorders) | 110 | 27 | 105
Toothache (Gastrointestinal disorders) | 11 | 5 | 10
Vomiting (Gastrointestinal disorders) | 61 | 41 | 70
Asthenia (General disorders) | 35 | 40 | 41
Chills (General disorders) | 11 | 1 | 14
Fatigue (General disorders) | 91 | 53 | 73
Influenza like illness (General disorders) | 9 | 3 | 16
Oedema peripheral (General disorders) | 76 | 23 | 66
Pyrexia (General disorders) | 56 | 23 | 57
Bronchitis (Infections and infestations) | 4 | 3 | 15
Influenza (Infections and infestations) | 6 | 7 | 12
Nasopharyngitis (Infections and infestations) | 33 | 14 | 38
Pneumonia (Infections and infestations) | 11 | 0 | 13
Sinusitis (Infections and infestations) | 14 | 4 | 17
Upper respiratory tract infection (Infections and infestations) | 16 | 7 | 28
Urinary tract infection (Infections and infestations) | 23 | 11 | 23
Alanine aminotransferase increased (Investigations) | 10 | 9 | 17
Aspartate aminotransferase increased (Investigations) | 12 | 11 | 28
Blood alkaline phosphatase increased (Investigations) | 12 | 11 | 25
Blood creatinine increased (Investigations) | 10 | 4 | 15
Haemoglobin decreased (Investigations) | 15 | 2 | 16
Weight decreased (Investigations) | 58 | 24 | 72
Decreased appetite (Metabolism and nutrition disorders) | 59 | 37 | 64
Dehydration (Metabolism and nutrition disorders) | 10 | 7 | 22
Diabetes mellitus (Metabolism and nutrition disorders) | 20 | 0 | 21
Hypercholesterolaemia (Metabolism and nutrition disorders) | 26 | 2 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 40 | 21 | 58
Hyperlipidaemia (Metabolism and nutrition disorders) | 16 | 2 | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 7 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 5 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 20 | 3 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 14 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 22 | 40
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 8 | 15
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 | 4 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 9 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 14 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 10 | 22
Dizziness (Nervous system disorders) | 24 | 16 | 18
Dysgeusia (Nervous system disorders) | 38 | 11 | 46
Headache (Nervous system disorders) | 62 | 30 | 52
Depression (Psychiatric disorders) | 14 | 3 | 18
Insomnia (Psychiatric disorders) | 28 | 17 | 27
Proteinuria (Renal and urinary disorders) | 10 | 2 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 21 | 54
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 13 | 34
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 44 | 3 | 38
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 12 | 29
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 2 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 21 | 0 | 17
Acne (Skin and subcutaneous tissue disorders) | 13 | 5 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 9 | 12
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 | 2 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 26 | 12 | 28
Erythema (Skin and subcutaneous tissue disorders) | 11 | 3 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 28 | 2 | 26
Onychoclasis (Skin and subcutaneous tissue disorders) | 14 | 2 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 40 | 26 | 42
Rash (Skin and subcutaneous tissue disorders) | 107 | 32 | 90
Flushing (Vascular disorders) | 4 | 6 | 12
Hypertension (Vascular disorders) | 24 | 9 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.